CLINICAL TRIAL: NCT03718481
Title: Perceptions of the Annual Review of Competence Progression (ARCP) in Surgical Training in the UK and Ireland: A Prospective Cross-Sectional Questionnaire Study.
Brief Title: Perceptions of the Annual Review of Competence Progression (ARCP) in Surgical Training in the UK and Ireland
Status: Completed | Type: Observational
Sponsor: University College Hospital Galway (Other)
Collaborators: The Association of Surgeons in Training (Other)
Responsible Party: Principal Investigator, Deirdre Nally, Research Fellow RCSI, ASiT representative for Republic of Ireland, University College Hospital Galway
Other Study IDs: ASiT ARCP
Record Dates: First submitted 2018-10-20; First posted 2018-10-24 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Education, Medical
Keywords: ARCP; Surgical Training; Assessment; Qualitative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Trainees: Trainee membership of the Association of Surgeons in Training (ASiT) in the UK and the Republic of Ireland
  Interventions: Other: ARCP Process

INTERVENTIONS:
Other: ARCP Process — One Annual Review of Competence Progression (ARCP) cycle. In the U.K., doctors, across all specialities, undergo an Annual Review of Competence Progression (ARCP) to evaluate performance during each training year and determine progression to the next year of training. Similar processes exist in the Republic of Ireland. The process and requirements for ARCP in the UK are specified in the Gold Guide, the Reference Guide for Postgraduate Specialty Training [1]. It defines ARCP as a formal process that uses evidence collected by trainees to review and record performance, demonstrate competencies achieved and inform decisions regarding progression in training

SUMMARY:
A Prospective Cross Sectional Questionnaire Study was conducted to evaluate surgical trainees' experiences of the ARCP process in order to identify areas for improvement.

DETAILED DESCRIPTION:
Background: Surgical trainees in the UK and Ireland undergo rigorous formative and summative assessments throughout each placement and appraisal at an Annual Review of Competence Progression (ARCP). The ARCP evaluates performance during each training year and determines progression to the next year of training. It is critical that the ARCP is a robust and fair process. The Association of Surgeons in Training (ASiT) sought to evaluate surgical trainees' experiences of the ARCP process in order to identify areas for improvement.

Methods: A Prospective Cross-Sectional Questionnaire Study was conducted An electronic survey was developed and distributed electronically to the trainee membership of ASiT in the UK and Republic of Ireland. A 57 point survey examined the specifics of one ARCP cycle as well as attitudes to the process in general. Quantitative analysis was performed, along with thematic analysis on the free-text comments.

ELIGIBILITY:
Inclusion Criteria:

* Must be a trainee member of ASiT
* All grades, Deaneries, including less than full-time/academic trainees are eligible for inclusion

Exclusion Criteria:

• Student members are excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgical Trainees in the UK and Ireland who are members of ASiT
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Experiences of Annual Review of Competence and Progression | Oct 2017-March 2018
  Experience of preparation, processes and standards. These will be measured on an anonymous, online survey (Survey monkey) and participants will be asked to rate their experiences of the ARCP using a likert scale. Specific experiences will include preparation for Annual Review of Competence and Progression-timing of decision making and value of the process as an educational tool and contribution of traineers, supervisors and the ARCP panel. Examples of questions are Did you feel your progression was fairly assessed? Possible answers include very fair, fair, neutral, not fair, very unfair

SECONDARY OUTCOMES:
Face to Face | Oct 2017- March 2018
  Trainees attitudes to a face to face Annual Review of Competence and Progression This will be measured on a likert scale similar to that outlined above (Strongly agree, agree, neutral, disagree, strongly disagree). There will be space for free text comments on the survey and a thematic analysis will be performed according to the steps of Braun and Clarke on the comments

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Nally, MCH, Principal Investigator — The Association of Surgeons in Training
Locations (1):
- Association of Surgeons in Training, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No